CLINICAL TRIAL: NCT03007602
Title: Effects of Upper Extremity Aerobic Exercise Training in Hematopoietic Stem Cell Transplantation Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gazi-231
Record Dates: First submitted 2016-12-16; First posted 2017-01-02 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Hematopoietic Stem Cell Transplantation; Aerobic Exercise
Keywords: Hematopoietic stem cell transplantation; Aerobic exercise; Quality of Life; Muscle Strength; Depression; exercise capacity; dyspnea; anxiety; fatigue; pulmonary functions
MeSH Terms: conditions — Depression; Dyspnea; Anxiety Disorders; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group: aerobic exercise (Experimental): The upper extremity aerobic exercise training with an arm ergometer will be performed in the treatment group so that training intensity will be between 60% and 80% of the maximum heart rate, dyspnea perception will be 3-4 according to Modified Borg Scale and fatigue perception will be 5-6 according to Modified Borg Scale, training duration will be a 6-week.
  Interventions: Other: Upper Extremity Aerobic Exercise
- Control group: deep breathing exercise (No Intervention): Deep breathing exercises combinated with arm movements will be given as a home schedule in the control group. Training duration will be a 6-week.

INTERVENTIONS:
Other: Upper Extremity Aerobic Exercise — Range of maximal heart rate is being followed by a polar band during supervised session each week.
  Aerobic exercise is being trained for 30 min-per/day, 3 days/week, 6 weeks. All sessions are being performed by a physiotherapist at cardiopulmonary rehabilitation department.
  Arms: Treatment group: aerobic exercise

SUMMARY:
Hematologic malignancy is a tumor of myeloid or lymphatic cells that affects lymph nodes with the involvement of blood, bone marrow or other organs.There are various treatment options for hematological malignancies ranging from follow-up to single or multiple agent chemotherapy, radiotherapy, immunotherapy and autologous or allogeneic hematopoietic stem cell transplantations (HSCT). The general recommendation for patients is to relax and avoid intense exercise, regardless of the devastating consequences of neglecting physical exercise. Patients also go to relaxation by reducing their activity to avoid fatigue, which leads to loss of muscle strength and endurance. As a consequence of all, fatigue, vomiting, weight loss, anemia, depression, decreased aerobic capacity, muscle weakness, decreased physical function and poor quality of life are observed in HSCT recipients. It has been shown that physical exercises improve oxygen consumption, depression and fatigue, cardiorespiratory fitness, muscle strength and physical well-being in patients with hematologic malignancies who are at stages of various treatments. In literature, effects of upper extremity aerobic exercise training have been investigated in patients with spinal cord injury, neuromuscular diseases, claudication, hypertension, multiple sclerosis, heart failure, paraplegic patients and healthy individuals. Results of these studies has shown that upper extremity aerobic exercise training improves walking distance, increases oxygen pulse, muscle strength and endurance of upper extremity. No study was observed to investigate the effects of upper extremity aerobic exercise training on exercise capacity and quality of life in HSCT recipients, as we know. For this reason, our aim is to investigate the effects of upper extremity aerobic exercise training on exercise capacity and quality of life in HSCT recipients.

DETAILED DESCRIPTION:
Minimum 30 allogeneic and autologous HSCT recipients (˃100 days past post-transplant status) will be included. Before and after 6-week upper extremity aerobic exercise training, maximal and submaximal exercise capacity, respiratory and peripheral muscle strength, pulmonary functions, physical activity, dyspnea and fatigue perception, anxiety, depression and quality of life were evaluated. Primary outcome measurements were exercise capacity and quality of life , secondary outcomes were respiratory and peripheral muscle strength, pulmonary functions, physical activity, dyspnea and fatigue perception, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* being an hematopoietic stem cell transplantation recipient during the intermediate/late post-transplant phase (>100 days),
* 18-65 years of age
* under standard medications.

Exclusion Criteria:

* having a cognitive disorder,
* orthopedic or neurological disease with a potential to affect functional capacity,
* comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute infections or pneumonia,
* problems which may prevent training such as visual problems and mucositis
* having metastasis to any region (bone etc.)
* having acute hemorrhage in the intracranial and / or lung and other areas
* having any contraindication to exercise training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
functional exercise capacity evaluation | 6-week
  Evaluated with 6-minute walking test

SECONDARY OUTCOMES:
pulmonary functions test | 6-week
  Evaluated with spirometer
muscle strength | 6-week
  Evaluated with a hand-held dynamometer for peripheral muscles, mouth pressure device for respiratory muscle strength
cough strength | 6-week
  Evaluated with peak flow meter
physical activity level | 6-week
  Evaluated with a metabolic holter
fatigue severity | 6-week
  Evaluated using Fatigue Severity Scale
anxiety and depression perception | 6-week
  Evaluated using Hospital Anxiety and Depression Scale
dyspnea perception | 6-week
  Evaluated using Modified Medical Research Council Dyspnea scale (MMRC) and Modified Borg Scale
quality of life level | 6-week
  evaluated using QOL using European Organization for Research and Treatment of Cancer QOL Questionnaire (EORTCQOL)
maximal exercise capacity evaluation | 6-week
  evaluated using Modified Incremental Shuttle Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, MSc., Study Chair — Gazi University; Meral Boşnak Güçlü, PhD., Study Director — Gazi University; Zübeyde Nur Özkurt, PhD., Principal Investigator — Gazi University; Münci Yağcı, PhD., Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- See also: 'Best supportive care' has had its day. — http://www.ncbi.nlm.nih.gov/pubmed/?term=2)%09Cullen+M.+%E2%80%99Best+supportive+care%E2%80%99+has+had+its+day.+The+Lancet+Oncology+2001%3B2(3)%3A173%E2%80%935.+%5BPUBMED%3A+11902569%5D
- See also: Management of bleeding and of invasive procedures in patients with platelet disorders and/or thrombocytopenia: Guidelines of the Italian Society for Haemostasis and Thrombosis (SISET). — http://www.ncbi.nlm.nih.gov/pubmed/?term=3)%09Tosetto+A%2C+Balduini+CL%2C+Cattaneo+M%2C+De+Candia+E%2C+Mariani+G%2C+Molinari+AC%2C+et+al.Management+of+bleeding+and+of+invasive+procedures+in+patients+with+platelet+disorders+and%2For+thrombocytopenia%3A+Guidelines+of+the+Italian+Society+for+Haemostasis+and+Thrombosis+(SISET).+Thrombosis+Research+2009%3B124(5)%3Ae13%E2%80%938.+%5BPUBMED%3A+19631969%5D
- See also: Aerobic physical exercise for adult patients with haematological malignancies. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Bergenthal+N%2C+Will+A%2C+Streckmann+F%2C+Wolkewitz+KD%2C+Monsef+I%2C+Engert+A%2C+Elter+T%2C+Skoetz+N.+Aerobic+physical+exercise+for+adult+patients+with+haematological+malignancies.+Cochrane+Database+Syst+Rev.